CLINICAL TRIAL: NCT05719857
Title: Diagnostic Role of the Hepatic Venous Pressure Gradient and Elastography in Porto-sinusoidal Vascular Disorder With Portal Hypertension
Brief Title: Hepatic Venous Pressure Gradient and Elastography in Porto-sinusoidal Vascular Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Guilherme Rezende, Associate Professor, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSVD-1
Record Dates: First submitted 2023-01-12; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Portal Hypertension; Non-Cirrhotic Portal Hypertension; Non-Cirrhotic Portal Fibrosis; Regenerative Nodular Hyperplasia; Incomplete Septal Cirrhosis; Obliterative Portal Venopathy; Idiopathic Non-Cirrhotic Portal Hypertension; Hepatoportal Sclerosis; Idiopathic Portal Hypertension; Vascular Disorder of Liver
MeSH Terms: conditions — Hypertension, Portal; Idiopathic Noncirrhotic Portal Hypertension | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: Comparative study between diagnostic methods, with a cross-sectional design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Portal hypertension patients with TE ≤ 20 kPa. (Experimental): All patients included will undergo HVPG measurement and US-guided percutaneous liver biopsy. The exams will be performed in sequence, in the laboratory of hepatic hemodynamics. Within 4 to 8 weeks, a multiparametric magnetic resonance imaging of the abdomen with elastography will be performed, concluding the protocol.
  Interventions: Procedure: Hepatic vein pressure gradient measurement; Procedure: Ultrasound-guided percutaneous liver biopsy; Diagnostic Test: Multiparametric Abdominal Magnetic Resonance with Elastography

INTERVENTIONS:
Procedure: Hepatic vein pressure gradient measurement — HVPG will be performed after light conscious sedation and with noninvasive vital sign monitoring. The right jugular vein will be catheterized with ultrasound assistance and after local anesthesia. Then a venous introducer will be placed and a balloon-tipped catheter will be advanced under fluoroscopic control into the right hepatic vein. Free hepatic pressure will be obtained with the balloon deflated, keeping the catheter tip in the right hepatic vein. Then, wedged venous pressure will be measured by inflating the balloon with 2 ml of air. At this moment, complete occlusion of the catheterized hepatic vein can be confirmed by injecting iodinated contrast and observing its retention. The presence of veno-venous communications can be detected during the test. To calculate the gradient, we perform the simple difference between the two measurements. Measurements will be performed in triplicate and the average used as the final value.
  Other Names: HVPG
Procedure: Ultrasound-guided percutaneous liver biopsy — Percutaneous liver biopsy will be performed with the aid of US to choose the best site for the procedure, minimizing the incidence of complications. With the patient in dorsal decubitus, venous analgesia with fentanyl 25-50 mcg will be performed. After marking the appropriate site, skin asepsis and antisepsis will be performed with Chlorhexidine® and topical anesthesia with 1% lidocaine. Then, the liver will be punctured using a 14G semi-automatic tru-cut single-use liver biopsy needle. The recovered material will be stored in a 50 ml flask with 10% formaldehyde. Patients will remain at rest supervised for 4 hours, with hourly measurement of blood pressure (BP), heart rate (HR) and assessment of symptoms (abdominal pain, nausea, etc.). In the absence of any complications, patients will be discharged from the hospital.
Diagnostic Test: Multiparametric Abdominal Magnetic Resonance with Elastography — The evaluation of the abdomen by MRI, with special interest to the liver and spleen, will be performed in a Siemens 3.0T Magnetom Prisma MR system. In addition to the routine protocol without contrast administration, MR elastography will be performed to assess liver stiffness and spleen stiffness. Data processing will be carried out at a Syngovia workstation.
  Other Names: MRE

SUMMARY:
Porto-sinusoidal vascular disorder (PSVD) is considered a rare cause of portal hypertension (PH), resulting from specific histological alterations that essentially affect the small portal branches and sinusoids, in the absence of cirrhosis.

In recent years, the recognition and importance of PSVD has increased, notably due to the widespread use of transient elastography (TE). However, the definitive diagnosis of PSVD can only be established through liver biopsy. Recent data show that PSVD should be suspected in patients with PH and TE ≤ 20 kPa and liver biopsy should be considered in this context.

The investigators hypothesize that hepatic venous pressure gradient (HVPG) and magnetic resonance liver elastography (MRE) may help in the selection of liver biopsy candidates for the diagnosis of PSVD.

The primary objective of the study is to describe HVPG and MRE values and liver biopsy findings in patients with PH and TE ≤ 20 kPa. The search for serum markers that can distinguish these patients from those with cirrhotic portal hypertension without the need for liver biopsy will also be the object of this study.

50 patients will be included, prospectively and retrospectively, in a comparative study between diagnostic methods, with a cross-sectional design.

DETAILED DESCRIPTION:
Porto-sinusoidal vascular disorder (PSVD) is considered a rare cause of portal hypertension (PH), resulting from specific histological alterations that essentially affect the small portal branches and sinusoids, in the absence of cirrhosis.

In recent years, the recognition and importance of PSVD has increased, notably due to the widespread use of transient elastography (TE). However, the definitive diagnosis of PSVD can only be established through liver biopsy. Recent data show that PSVD should be suspected in patients with PH and TE ≤ 20 kPa and liver biopsy should be considered in this context.

The investigators hypothesize that hepatic venous pressure gradient (HVPG) and magnetic resonance liver elastography (MRE) may help in the selection of liver biopsy candidates for the diagnosis of PSVD.

Primary objectives are:

* To describe the measurement of the hepatic venous pressure gradient (in mmHg) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
* To describe hepatic (in kPa) and splenic (in kPa) stiffness measured by magnetic resonance elastography in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
* To describe the frequency of major histological findings for the diagnosis of portal sinusoidal vascular disorder (obliterative portal venopathy, regenerative nodular hyperplasia and incomplete septal cirrhosis) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.

Secondary objectives are:

* To describe the frequency of hepatic vein-to-vein communications in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
* To describe the frequency of minor histological findings for the diagnosis of portal sinusoidal vascular disease (portal tract abnormalities, architectural disturbances, nonzonal sinusoidal dilatation, mild perisinusoidal fibrosis) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
* To compare the serum values of von Willebrand antigen factor (IU/mL) between patients diagnosed with porto-sinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.
* To compare the serum titers of procollagen III amino-terminal peptide (mcg/l) between patients diagnosed with portosinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.
* To compare the serum titers of anti-endothelial cell antibodies between patients diagnosed with portosinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.

  50 patients will be included, prospectively and retrospectively, in a comparative study between diagnostic methods, with a cross-sectional design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with specific signs of portal hypertension:

  1. Endoscopic: esophagogastric/ectopic varices;
  2. On imaging (US, CT or MRI): portosystemic collateral veins;
* Transient hepatic elastography with valid values ≤ 20 kPa;
* Signed written informed consent form.

Exclusion Criteria:

* Contraindications to HVPG or percutaneous liver biopsy:

  1. Pregnancy
  2. Allergy to iodine
  3. Chronic kidney disease with creatinine clearance < 50 ml/min
  4. Anticoagulation
  5. RNI > 1.5
  6. Platelets < 50,000/mm3
* Confounding factors:

  1. Hepatitis C treated with SVR
* Conditions that exclude the diagnosis of PSVD:

  1. History of bone marrow transplant
  2. Budd-Chiari
  3. Congestive heart failure or Fontan surgery
  4. Abernethy's Syndrome
  5. Hereditary hemorrhagic telangiectasia
  6. Chronic cholestatic diseases
  7. Neoplastic hepatic infiltration
  8. Sarcoidosis
  9. Congenital hepatic fibrosis
  10. Hepatosplenic schistosomiasis
  11. Portal cavernoma / thrombosis with complete occlusion of the main portal vein.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Hepatic venous pressure gradient measurement | 12 months
  To describe the measurement of the hepatic venous pressure gradient (in mmHg) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
Magnetic resonance elastography | 12 months
  To describe hepatic (in kPa) and splenic (in kPa) stiffness measured by magnetic resonance elastography in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
Liver biopsy major findings | 12 months
  To describe the frequency of major histological findings for the diagnosis of portal sinusoidal vascular disorder (obliterative portal venopathy, regenerative nodular hyperplasia and incomplete septal cirrhosis) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.

SECONDARY OUTCOMES:
Hepatic vein-to-vein communications | 12 months
  To describe the frequency of hepatic vein-to-vein communications in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
Liver biopsy minor findings | 12 months
  To describe the frequency of minor histological findings for the diagnosis of portal sinusoidal vascular disease (portal tract abnormalities, architectural disturbances, nonzonal sinusoidal dilatation, mild perisinusoidal fibrosis) in patients with portal hypertension and transient hepatic elastography ≤ 20 kPa.
Non-invasive markers - von Willebrand antigen factor | 12 months
  To compare the serum values of von Willebrand antigen factor (IU/mL) between patients diagnosed with porto-sinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.
Non-invasive markers - procollagen III amino-terminal peptide | 12 months
  To compare the serum titers of procollagen III amino-terminal peptide (mcg/l) between patients diagnosed with portosinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.
Non-invasive markers - anti-endothelial cell antibodies | 12 months
  To compare the serum titers of anti-endothelial cell antibodies between patients diagnosed with portosinusoidal vascular disorder and those diagnosed with cirrhosis, after analysis of liver biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme FM Rezende, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Hospital Universitário Clementino Fraga Filho / Universidade Federal do Rio de Janeiro (UFRJ), Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huwart L, Sempoux C, Vicaut E, Salameh N, Annet L, Danse E, Peeters F, ter Beek LC, Rahier J, Sinkus R, Horsmans Y, Van Beers BE. Magnetic resonance elastography for the noninvasive staging of liver fibrosis. Gastroenterology. 2008 Jul;135(1):32-40. doi: 10.1053/j.gastro.2008.03.076. Epub 2008 Apr 4. PMID 18471441
- [Background] Berzigotti A, Seijo S, Reverter E, Bosch J. Assessing portal hypertension in liver diseases. Expert Rev Gastroenterol Hepatol. 2013 Feb;7(2):141-55. doi: 10.1586/egh.12.83. PMID 23363263
- [Background] Cerda Reyes E, Gonzalez-Navarro EA, Magaz M, Munoz-Sanchez G, Diaz A, Silva-Junior G, Triguero A, Lafoz E, Camprecios G, Orts L, Perez-Campuzano V, Seijo S, Rubio L, Turon F, Baiges A, Hernandez-Gea V, Alvarez-Larran A, Juan M, Garcia-Pagan JC. Autoimmune biomarkers in porto-sinusoidal vascular disease: Potential role in its diagnosis and pathophysiology. Liver Int. 2021 Sep;41(9):2171-2178. doi: 10.1111/liv.14997. Epub 2021 Jul 11. PMID 34173316
- [Background] D'Amico G, Garcia-Tsao G, Pagliaro L. Natural history and prognostic indicators of survival in cirrhosis: a systematic review of 118 studies. J Hepatol. 2006 Jan;44(1):217-31. doi: 10.1016/j.jhep.2005.10.013. Epub 2005 Nov 9. No abstract available. PMID 16298014
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] De Gottardi A, Rautou PE, Schouten J, Rubbia-Brandt L, Leebeek F, Trebicka J, Murad SD, Vilgrain V, Hernandez-Gea V, Nery F, Plessier A, Berzigotti A, Bioulac-Sage P, Primignani M, Semela D, Elkrief L, Bedossa P, Valla D, Garcia-Pagan JC; VALDIG group. Porto-sinusoidal vascular disease: proposal and description of a novel entity. Lancet Gastroenterol Hepatol. 2019 May;4(5):399-411. doi: 10.1016/S2468-1253(19)30047-0. PMID 30957754
- [Background] Elkrief L, Lazareth M, Chevret S, Paradis V, Magaz M, Blaise L, Rubbia-Brandt L, Moga L, Durand F, Payance A, Plessier A, Chaffaut C, Valla D, Malphettes M, Diaz A, Nault JC, Nahon P, Audureau E, Ratziu V, Castera L, Garcia Pagan JC, Ganne-Carrie N, Rautou PE; ANRS CO12 CirVir Group. Liver Stiffness by Transient Elastography to Detect Porto-Sinusoidal Vascular Liver Disease With Portal Hypertension. Hepatology. 2021 Jul;74(1):364-378. doi: 10.1002/hep.31688. Epub 2021 Jun 11. PMID 33345307
- [Background] European Association for Study of Liver; Asociacion Latinoamericana para el Estudio del Higado. EASL-ALEH Clinical Practice Guidelines: Non-invasive tests for evaluation of liver disease severity and prognosis. J Hepatol. 2015 Jul;63(1):237-64. doi: 10.1016/j.jhep.2015.04.006. Epub 2015 Apr 21. No abstract available. PMID 25911335
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on non-invasive tests for evaluation of liver disease severity and prognosis - 2021 update. J Hepatol. 2021 Sep;75(3):659-689. doi: 10.1016/j.jhep.2021.05.025. Epub 2021 Jun 21. PMID 34166721
- [Background] Ferlitsch M, Reiberger T, Hoke M, Salzl P, Schwengerer B, Ulbrich G, Payer BA, Trauner M, Peck-Radosavljevic M, Ferlitsch A. von Willebrand factor as new noninvasive predictor of portal hypertension, decompensation and mortality in patients with liver cirrhosis. Hepatology. 2012 Oct;56(4):1439-47. doi: 10.1002/hep.25806. Epub 2012 Aug 27. PMID 22532296
- [Background] Goel A, Ramakrishna B, Muliyil J, Madhu K, Sajith KG, Zachariah U, Ramachandran J, Keshava SN, Selvakumar R, Chandy GM, Elias E, Eapen CE. Use of serum vitamin B12 level as a marker to differentiate idiopathic noncirrhotic intrahepatic portal hypertension from cryptogenic cirrhosis. Dig Dis Sci. 2013 Jan;58(1):179-87. doi: 10.1007/s10620-012-2361-7. Epub 2012 Aug 24. PMID 22918688
- [Background] Gronbaek H, Sandahl TD, Mortensen C, Vilstrup H, Moller HJ, Moller S. Soluble CD163, a marker of Kupffer cell activation, is related to portal hypertension in patients with liver cirrhosis. Aliment Pharmacol Ther. 2012 Jul;36(2):173-80. doi: 10.1111/j.1365-2036.2012.05134.x. Epub 2012 May 16. PMID 22591184
- [Background] Khanna R, Sarin SK. Noncirrhotic Portal Hypertension: Current and Emerging Perspectives. Clin Liver Dis. 2019 Nov;23(4):781-807. doi: 10.1016/j.cld.2019.07.006. PMID 31563222
- [Background] La Mura V, Reverter JC, Flores-Arroyo A, Raffa S, Reverter E, Seijo S, Abraldes JG, Bosch J, Garcia-Pagan JC. Von Willebrand factor levels predict clinical outcome in patients with cirrhosis and portal hypertension. Gut. 2011 Aug;60(8):1133-8. doi: 10.1136/gut.2010.235689. Epub 2011 Mar 22. PMID 21427197
- [Background] Morikawa H, Tamori A, Nishiguchi S, Enomoto M, Habu D, Kawada N, Shiomi S. Expression of connective tissue growth factor in the human liver with idiopathic portal hypertension. Mol Med. 2007 May-Jun;13(5-6):240-5. doi: 10.2119/2006-00093.Morikawa. PMID 17622321
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Seijo S, Reverter E, Miquel R, Berzigotti A, Abraldes JG, Bosch J, Garcia-Pagan JC. Role of hepatic vein catheterisation and transient elastography in the diagnosis of idiopathic portal hypertension. Dig Liver Dis. 2012 Oct;44(10):855-60. doi: 10.1016/j.dld.2012.05.005. Epub 2012 Jun 19. PMID 22721839
- [Background] Sharma P, Agarwal R, Dhawan S, Bansal N, Singla V, Kumar A, Arora A. Transient Elastography (Fibroscan) in Patients with Non-cirrhotic Portal Fibrosis. J Clin Exp Hepatol. 2017 Sep;7(3):230-234. doi: 10.1016/j.jceh.2017.03.002. Epub 2017 Mar 14. PMID 28970710
- [Background] Siramolpiwat S, Seijo S, Miquel R, Berzigotti A, Garcia-Criado A, Darnell A, Turon F, Hernandez-Gea V, Bosch J, Garcia-Pagan JC. Idiopathic portal hypertension: natural history and long-term outcome. Hepatology. 2014 Jun;59(6):2276-85. doi: 10.1002/hep.26904. Epub 2014 Feb 28. PMID 24155091
- [Background] Waidmann O, Brunner F, Herrmann E, Zeuzem S, Piiper A, Kronenberger B. Macrophage activation is a prognostic parameter for variceal bleeding and overall survival in patients with liver cirrhosis. J Hepatol. 2013 May;58(5):956-61. doi: 10.1016/j.jhep.2013.01.005. Epub 2013 Jan 16. PMID 23333526